CLINICAL TRIAL: NCT06639022
Title: Comparison of the Postoperative Analgesic Efficacy of Serratus Posterior Superior Intercostal Plane Block and Erector Spinae Plane Block in Anterior Cervical Discectomy
Brief Title: Comparison of the Postoperative Analgesic Efficacy of SPSIPB and ESPB in Anterior Cervical Discectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Atakan Sezgi, Principal İnvestigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEŞH-EK1-2024-0126
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Anterior Cervical Discectomy; Peripheral Nerve Block; Pain Management
Keywords: Anterior Cervical Discectomy; Serratus Posterior Superior Intercostal Plane Block; Erector Spinae Plane Block
MeSH Terms: conditions — Agnosia | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Serratus posterior superior intercostal plane block (Active Comparator): After the patients are monitored and in the supine position, after appropriate field sterilization, a serratus posterior superior intercostal plane block will be performed on the patients using 30 ml of local anesthetic solution (0.25% bupivacain) under ultrasound guidance. In the intraoperative period, intravenous analgesics (dexketoprofen 50 mg, tramadol 100 mg) will be given.
  Interventions: Procedure: Serratus posterior superior intercostal plane block
- Erector spinae plane block (Active Comparator): After the patients are monitored and in the supine position, after appropriate field sterilization, a erector spinae plane block will be performed on the patients using 30 ml of local anesthetic solution (0.25% bupivacain) under ultrasound guidance. In the intraoperative period, intravenous analgesics (dexketoprofen 50 mg, tramadol 100 mg) will be given.
  Interventions: Procedure: Erector spinae plane block
- Group without peripheral nerve block (Active Comparator): After the patients are monitored, they will be operated under general anesthesia without peripheral nerve block and intraoperative intravenous analgesics (dexketoprofen 50 mg, tramadol 100 mg) will be given.
  Interventions: Procedure: Group without peripheral nerve block

INTERVENTIONS:
Procedure: Serratus posterior superior intercostal plane block — Serratus posterior superior intercostal plane block will be performed on the patients using 30 ml of 0.25% bupivacaine under ultrasound guidance.
  Additionally, in the postoperative period a paracetamol dose of 1 g every 8 hours and a dexketoprofen dose of 50 mg twice daily were administered iv for multimodal analgesia.
  Arms: Serratus posterior superior intercostal plane block
Procedure: Erector spinae plane block — Erector spinae plane block will be performed on the patients using 30 ml of 0.25% bupivacaine under ultrasound guidance.
  Additionally, in the postoperative period a paracetamol dose of 1 g every 8 hours and a dexketoprofen dose of 50 mg twice daily were administered iv for multimodal analgesia.
  Arms: Erector spinae plane block
Procedure: Group without peripheral nerve block — In the postoperative period a paracetamol dose of 1 g every 8 hours and a dexketoprofen dose of 50 mg twice daily were administered iv for multimodal analgesia.
  Arms: Group without peripheral nerve block

SUMMARY:
Anterior cervical discectomy is an operation performed for complaints of pain, numbness or loss of strength due to cervical disc disease. With this operation, pressure due to herniation on the upper neck area, spinal cord or nerve roots is relieved. It is performed by microscopic method from the front of the neck.

Nerve blocks reduces opioid consumption in the postoperative period by providing better pain control and therefore has advantages such as fewer side effects and less risk of pulmonary and cardiac complications.

In this study; it was aimed to compare the analgesic effectiveness of serratus posterior superior intercostal plane block and erector spinae plane block, with each other and with the control group in the postoperative period in patients who underwent anterior cervical discectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* American Society of Anesthesiologists (ASA) score I-II-III
* Body Mass Index (BMI) between 18-30 kg/m2

Exclusion Criteria:

* Patients under 18 and over 80 years of age
* ASA score IV and above
* Patients with a history of bleeding diathesis
* BMI below 18 or above 30 kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | On the operation day
  Pain will be assessed at rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at 0st, 1st, 2nd,4th, 12th, and 24th hours after surgery.

SECONDARY OUTCOMES:
Intraoperative remifentanil consumption Intraoperative opioid consumption | Intraoperative period
  Remifentanil consumption for intraoperative period will be recorded
Postoperative Tramadol Consumption | On the operation day
  Tramadol consumption for 24 hours will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Altındağ, Ankara, Turkey (Türkiye)